CLINICAL TRIAL: NCT01449513
Title: A Phase 1, Two-stage, Single-centre, Open Label, Within- and Between-subject Comparison Trial to Explore the Biological Effects of PEP005 (Ingenol Mebutate) Gel, 0.05%, Applied Once Daily for 2 Consecutive Days in Subjects With Actinic Keratosis on the Upper Extrem-ity. A Single-arm First Stage Followed by a Two-arm, Parallel Group, Randomized, Placebo (Vehicle) -Controlled Second Stage
Brief Title: PEP005 Gel - Biological Effects in Actinic Keratosis Assessed by Reflectance Confocal Microscopy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LP0041-03
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2016-04

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 Gel 0.05% (Active Comparator): active ingredient of PEP005: Ingenol mebutate
  Interventions: Drug: Ingenol mebutate
- Placebo Gel (Placebo Comparator): Vehicle of PEP005 Gel
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Ingenol mebutate — 0.05% Ingenol mebutate Gel once daily for 2 consecutive days
  Other Names: PEP005
  Arms: PEP005 Gel 0.05%
Drug: Placebo Gel — Gel vehicle of PEP005
  Arms: Placebo Gel

SUMMARY:
This trial will be conducted to explore the biological effects in the skin following treatment with PEP005 Gel, 0.05% administered for two consecutive days, assessed by reflectance confocal microscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age
2. Subjects with AK lesions and subclinical AK lesions within a contiguous 25 cm2 area on the upper extremity
3. Subjects must have a 25 cm2 area of normal skin on the inner upper arm
4. Female subjects must be of either:• Non-childbearing potential, post-menopausal, or have a confirmed clinical history of sterility or • Childbearing potential, with a confirmed negative urine pregnancy test prior to exposure.
5. Female subjects of childbearing potential must be willing to consent to using high effective methods of contraception
6. Ability to follow trial instructions and likely to complete all trial requirements
7. Obtained written informed consent prior to any trial-related procedures

Exclusion Criteria:

1. Location of the selected treatment areas:• Within 5 cm of an incompletely healed wound or infected area of the skin • Within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma(SCC)
2. History or evidence of skin conditions other than the trial indication that would interfere with evaluation of the investigational product
3. Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a significant AE or interfere with assessments of safety during the course of the trial, as determined by Investigator clinical judgment
4. Anticipated need for in-patient hospitalisation or in-patient surgery during the trial period.
5. Current participation in any other interventional clinical trial
6. Subjects who have received treatment with any non-marketed drug product within the last two months
7. Previous enrolment in this clinical trial
8. Prohibited Therapies and/or Medications 2 weeks prior to the Screening visit within 2 cm of selected treatment area:•Cosmetic or therapeutic procedures •Use of acid-containing therapeutic products • Use of topical salves or topical steroids
9. Prohibited Therapies and/or Medications: within 4 weeks prior to the Screening visit: • Treatment with immunomodulators, cytotoxic drugs or interferon/interferon inducers,systemic medications that suppress the immune system, or with UVB
10. Prohibited Therapies and/or Medications: within 8 weeks prior to the Screening visit: • Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 2 cm of the selected treatment areas.
11. Use of systemic retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eggert Stockfleth, Prof Dr med, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date: 27-Sep-2011 (FSFV - first subject first visit) Completion date: 22-May-2012 (LSLV - last subject last visit)
Groups:
- Ingenol Mebutate Gel (PEP005 Gel): Ingenol mebutate gel (PEP005 gel)
  Ingenol mebutate gel (0.05%) once daily on two consecutive days to an 25cm2 area
- Vehicle: Vehicle of PEP005 Gel
  Vehicle gel once daily on two consecutive days to an 25cm2 area
Period: Overall Study
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Started | 16 | 8
Completed | 16 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (7.5) | 69.9 (3.5) | 70.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Germany | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by Reflectance Confocal Microscopy (RCM) in actinic keratosis (AK) skin.This RCM imaging technique is a relatively new non-invasive, real-time evaluation method to generate horizontal skin sections at a resolution comparable to routine histology.
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 2
Population: As stated in the outcome measure, the degree of infiltration will be assessed for subjects receiving Ingenol Mebutate Gel. Therefor this is 0 for all subjects receiving vehicle.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage change | 1.42 (0.94) |

2. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by Reflectance Confocal Microscopy (RCM) in Sub actinic keratosis (AK) skin.
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 1.52 (0.74) |

3. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in normal skin.
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.94 (0.68) |

4. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in AK (actinic keratosis) skin
Time Frame: Baseline to Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 2.24 (0.77) |

5. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in Sub AK (actinic keratosis) skin.
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 2.07 (0.76) |

6. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in normal skin
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 1.38 (0.50) |

7. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in AK (actinic keratosis) skin
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.90 (0.90) |

8. Primary Outcome: Change in Degree of Infiltration
Description: Change from baseline in the degree of infiltration of the epidermis by inflammatory cells following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in Sub AK (actinic keratosis) skin
  The degree of infiltration of the epidermis by inflammatory cells will be based on "inflammation/small bright cells" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel. The degree of infiltration of the dermis by inflammatory cells will be based on "inflammatory cells in the dermis" (grading 0-3) as assessed by RCM from baseline across the trial period for the subjects receiving PEP005 Gel.
Time Frame: Baseline to Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 1.16 (0.95) |

9. Primary Outcome: Change in Degree of Infiltration
Description: as for outcome 6
Time Frame: Baseline to Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.31 (0.60) |

10. Primary Outcome: Change in Degree of Infiltration
Description: as for outcome 7
Time Frame: Baseline to Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | -0.60 (0.62) |

11. Primary Outcome: Change in Degree of Infiltration
Description: as for outcome 8
Time Frame: Baseline to Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.03 (0.47) |

12. Primary Outcome: Change in Degree of Infiltration
Description: as for outcome 6
Time Frame: Baseline to Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0 (0) |

13. Primary Outcome: Change in Degree of Necrosis
Description: Change from baseline in the degree of necrosis in the epidermis following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in AK (actinic keratosis) skin
Time Frame: Baseline to Day 2
Population: As stated in the outcome measure, the degree of necrosis will be assessed for subjects receiving Ingenol Mebutate Gel. Therefor this is 0 for all subjects receiving vehicle.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 1.69 (0.93) |

14. Primary Outcome: Change in Degree of Necrosis
Description: Change from baseline in the degree of necrosis in the epidermis following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in Sub AK (actinic keratosis) skin
Time Frame: Baseline to Day 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 1.42 (0.90) |

15. Primary Outcome: Change in Degree of Necrosis
Description: Change from baseline in the degree of necrosis in the epidermis following treatment with ingenol mebutate gel, 0.05% as assessed by RCM (Reflectance Confocal Microscopy) in normal skin
Time Frame: Baseline to Day 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.81 (0.66) |

16. Primary Outcome: Change in Degree of Necrosis
Description: Change from baseline in the degree of necrosis in the epidermis following treatment with ingenol mebutate gel, 0.05% as assessed by RCM(Reflectance Confocal Microscopy) in AK (actinic keratosis) skin
Time Frame: Baseline to Day 3
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 2.44 (0.69) |

17. Primary Outcome: Change in Degree of Necrosis
Description: as for outcome 14
Time Frame: Baseline to Day 3
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 2.16 (0.86) |

18. Primary Outcome: Change in Degree of Necrosis
Description: as for outcome 15
Time Frame: Baseline to Day 3
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 1.38 (0.72) |

19. Primary Outcome: Change in Degree of Necrosis
Description: as for outcome 13
Time Frame: Baseline to Day 8
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.31 (0.66) |

20. Primary Outcome: Change in Degree of Necrosis
Description: as for outcome 14
Time Frame: Baseline to Day 8
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0.28 (0.68) |

21. Primary Outcome: Change in Degree of Necrosis
Description: Change from baseline in the degree of necrosis in the epidermis following treatment with ingenol mebutate gel,0.05% as assessed by RCM (Reflectance Confocal Microscopy) in normal skin
Time Frame: Baseline to Day 8
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0 (0) |

22. Primary Outcome: Change in Degree of Necrosis
Description: as for outcome 13
Time Frame: Baseline to Day 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0 (0) |

23. Primary Outcome: Change in Degree of Necrosis
Description: as for outcome 14
Time Frame: Baseline to Day 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0 (0) |

24. Primary Outcome: Change in Degree of Necrosis
Description: Change from baseline in the degree of necrosis in the epidermis following treatment with ingenol mebutate gel, 0.05% as assessed by RCM in normal skin
Time Frame: Baseline to Day 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Number analyzed (Participants) | 16 | 0
percentage of change | 0 (0) |

ADVERSE EVENTS:
Arm/Group | Ingenol Mebutate Gel (PEP005 Gel) | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/8
Other Adverse Events (participants affected / at risk) | 16/16 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Mebutate Gel (PEP005 Gel) (N=16) | Vehicle (N=8)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol Mebutate Gel (PEP005 Gel) (N=16) | Vehicle (N=8)
Angina pectoris (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Pain (General disorders) | 10 | 0
Swelling (General disorders) | 1 | 0
Postoperative wound (Infections and infestations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 8 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.